CLINICAL TRIAL: NCT01606124
Title: Randomized Phase II Trial of Polyphenon E vs.Placebo in Patients at High Risk of Recurrent Colonic Neoplasia
Brief Title: Polyphenon E in Treating Patients With High-Risk of Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: pending expiration of the supply of study agent.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC084C; NCI-2012-00058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT01974960 (obsolete NCT alias)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-05

CONDITIONS: Advanced Colorectal Adenomas; Adenocarcinoma of the Colon; Stage I Colon Cancer; Stage II Colon Cancer; Stage III Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Green Tea Catechin Extract) (Experimental): Patients receive Polyphenon E PO BID. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: defined green tea catechin extract; Other: questionnaire administration; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: questionnaire administration; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: defined green tea catechin extract — Given PO
  Other Names: Polyphenon E
  Arms: Arm I (Green Tea Catechin Extract)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well Polyphenon E works in treating patients with high-risk of colorectal cancer. Polyphenon E contains ingredients that may prevent or slow colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine whether POLYE (Polyphenon E) treatment is associated with a significant percent decrease in the number of rectal Aberrant Crypt Foci (ACF) (% change in ACF) identified during the pre-intervention and post-intervention chromoendoscopy exams. SECONDARY OBJECTIVES: I. To determine the relative tolerability and safety of treatment with 2 capsules of POLYE taken twice a day by mouth (Note: each capsule of Polyphenon E contains approximately 200 mg of epigallocatechin gallate (EGCG) versus placebo administered for 6 months. TERTIARY OBJECTIVES: I. To determine the effect of the study drug vs. placebo on EGCG levels in plasma and to correlate EGCG levels with drug compliance and toxicity. II. To characterize ACF based on four criteria and correlate such characterizations with the intervention (vs placebo), as well as exploring the natural history of ACF over 6 months in persons at high risk for colorectal cancer randomized to placebo. III. To correlate the 6-month measurements of ACF size (e.g., number of crypts/ACF), number, morphology, and histopathology with the adenoma recurrence data at the next surveillance endoscopy. IV. To assess caffeine and black tea consumption via a Beverage Consumption Questionnaire and correlate with study endpoints. V. To assess the effects of POLYE versus placebo on a focused panel of tissue biomarkers using re- and post-intervention biopsy samples obtained from ACF and normal-appearing rectal mucosa. Residual tissue will be stored for further analysis. VI. To study the association of clinical (toxicity and/or ACF response or activity) with the pharmacokinetic parameters, and/or biologic (pharmacodynamic) results. OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive Polyphenon E orally (PO) twice daily (BID). ARM II: Patients receive placebo PO BID. Courses in both arms repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Current or prior advanced adenomas. Participants with advanced adenomas are defined as participants who have polyps >= 1 cm, who have tubulovillous adenomas (25-75 percent villous features), who have villous adenomas (>75 percent villous), or who have severe dysplasia
* Prior curatively resected Tumor, Node, Metastasis (TNM) stage II and III colon cancer >= 3 years out from treatment by surgery with/without adjuvant chemotherapy; NOTE: patients with stage I (T1,2 N0) colon cancer treated by endoscopic or surgical therapy are eligible at anytime after such therapy; patients with prior stage IV disease must be >= 5 years status post surgical resection of all metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to discontinue regular usage of calcium supplements; Exception: multi-vitamin; regular use defined as a frequency of 7 consecutive days for > 3 weeks
* Willingness to provide mandatory tissue and blood for protocol specified research; residual tissue and/or blood may be used for future research Negative pregnancy test =< 7 days prior to registration/randomization
* Hemoglobin (Hgb) >= 12.0 g/dL (women), >= 13.5 g/dL (men) at Mayo Clinic or within normal limits at an outside laboratory
* Platelet count >= 100,000/ul
* White blood cells (WBC) >= 3,000/ul
* Alanine aminotransferase (ALT) within institutional limits of normal
* Alkaline phosphatase within institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) within institutional limits of normal
* Total bilirubin within institutional limits of normal
* Serum calcium =< institutional ULN
* Serum creatinine =< 1.5 x institutional ULN
* >= 5 rectal ACF detected by chromoendoscopy =< 45 days prior to registration/randomization
* Endoscopy =< 45 days prior to registration/randomization; Note: All adenomas or polyps will be removed according to institutional standards of care, and the cecum must visualized; this may be done at the same time as the chromoendoscopy

Exclusion Criteria:

* Any history of rectal cancer; Exception: transanal excision without radiation
* Known diagnosis of colon heritable cancer syndrome (Familial adenomatous polyposis [FAP], hereditary nonpolyposis colorectal cancer [HNPCC]) or inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Inability to swallow capsules
* Bleeding diathesis
* Any invasive malignancy =< 5 years prior to pre-registration;

  * Exceptions:
  * patients with nonmelanoma skin cancers that were treated with simple excisional biopsy or stage I (T1,2 N0)
  * colon cancer treated by endoscopic therapy or surgery are eligible
* History of gastroduodenal ulcers documented =< 1 year
* Known inability to participate in the scheduled follow-up tests
* Significant medical or psychiatric problems which would make the participant a poor protocol candidate, in the opinion of the treating physician
* Total colectomy
* Colostomy
* History of pelvic or rectal radiation therapy
* History of liver disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Concomitant corticosteroids or anticoagulants needed on a regular or predictable intermittent basis
* Use of non-study investigational agent(s) =< 3 months prior to preregistration
* Chemotherapy =< 6 months prior to pre-registration; Note: Topical chemotherapy will be assessed on a case-by-case basis
* Any of the following: * Pregnant women * Nursing women * Men or women of childbearing potential who are unwilling to employ adequate contraception Note: This study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown
* Over-the-counter green tea or green tea extract use =< 6 weeks prior to pre-registration; consumption of over the counter green tea extracts or drinking of green tea is not permitted during the treatment portion of this trial
* Regular use of nonsteroidal anti-inflammatory drugs (NSAIDs) =< 6 weeks prior to pre-registration; regular use of NSAIDs is defined as a frequency of 7 consecutive days (1 week) for > 3 weeks; participant must abstain from regular use of NSAIDs for the duration of the study; Exception: low dose aspirin (81 mg) for those participants who are chronic users of aspirin prior to the beginning of the study
* Use of non-study investigational agents while on study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05-21 (Actual); Study Completion 2015-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sinicrope, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of Illinois, Chicago, Illinois
  - Hines Veteran's Administration Hospital, Hines, Illinois
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was closed to accrual early due to a pending expiration of the supply of study agent.
Groups:
- Arm I (Polyphenon E): Patients receive two capsules Polyphenon E (each capsule of Polyphenon E contains approximately 200 mg epigallocatechin gallate (EGCG)) PO BID. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
- Arm II (Placebo): Patients receive two capsules placebo PO BID. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Polyphenon E) | Arm II (Placebo)
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Polyphenon E) | Arm II (Placebo) | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (17.0) | 61.4 (7.9) | 59.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 13 | 12 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Rectal ACF, Pre- and Post Intervention at 6 Months
Description: The primary endpoint is based on a modified intent-to-treat procedure which includes all patients with baseline and 6-month ACF data. The percent change in rectal ACF (≤ 15 cm from the anal verge) for each patient is calculated as their Pre-Registration number of rectal ACF minus the number of rectal ACF present at the 6-month post-intervention exam, divided by the number of rectal ACF present at Pre-Registration times 100.
Time Frame: 6 months
Population: Patients with baseline and 6-month ACF data were included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Arm I (Polyphenon E) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 17
percentage change | 3.7 (49.1) | 0.0 (62.7)
Statistical Analysis 1: Comparison: Arm I (Polyphenon E) vs Arm II (Placebo); Test type: Superiority; p = 0.5631, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Tolerability as Estimated Using the Percent Dose of Treatment Received at 6 Months
Description: Tolerability as estimated using the percent dose of treatment received for each patient by dividing the total dose received by the targeted (i.e., protocol specified) total dose.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of targeted dose
Arm/Group | Arm I (Polyphenon E) | Arm II (Placebo)
Number analyzed (Participants) | 19 | 20
percentage of targeted dose | 83.2 (29.3) | 91.7 (24.0)
Statistical Analysis 1: Comparison: Arm I (Polyphenon E) vs Arm II (Placebo); Test type: Superiority; p = 0.1439, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Arm I (Polyphenon E) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 4/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Polyphenon E) (N=19) | Arm II (Placebo) (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (6)
Fatigue (General disorders) | 0 (0) | 1 (6)
Flu like symptoms (General disorders) | 0 (0) | 1 (6)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (6)
Dizziness (Nervous system disorders) | 0 (0) | 1 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes